CLINICAL TRIAL: NCT00105456
Title: registHER: An Observational Cohort Study of Patients With HER2 Positive Metastatic Breast Cancer
Brief Title: A Study of Patients With HER2-Positive Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Other Study IDs: H2757n
Record Dates: First submitted 2005-03-14; First posted 2005-03-15 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2010-05

CONDITIONS: Breast Cancer
Keywords: HER2-Positive Metastatic Breast Cancer; HER2
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is a prospective observational cohort study designed to describe effectiveness and safety (treatment outcomes and clinically significant cardiac adverse events, respectively) in patients with HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent document (unless the IRB has granted a waiver of consent)
* Signed Authorization for the Use and Disclosure of Health Information document
* HER2-positive breast cancer
* Initial diagnosis of metastatic (Stage IV) breast cancer within 6 months prior to enrollment
* Availability of cancer-specific historical data points in the patient's medical records

Exclusion Criteria:

* There are no exclusion criteria for participation in this trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from managed care organizations, community physicians or practices, and academic centers.
Sampling Method: Non-Probability Sample
Enrollment: 1000
Dates: Start 2003-03; Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isaiah Dimery, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Yardley DA, Tripathy D, Brufsky AM, Rugo HS, Kaufman PA, Mayer M, Magidson J, Yoo B, Quah C, Ulcickas Yood M. Long-term survivor characteristics in HER2-positive metastatic breast cancer from registHER. Br J Cancer. 2014 May 27;110(11):2756-64. doi: 10.1038/bjc.2014.174. Epub 2014 Apr 17. PMID 24743708